CLINICAL TRIAL: NCT07265960
Title: Effect of Virtual Reality and Stress Ball Interventions on Procedure-Related Fear, Pain, Anxiety, and Patient Satisfaction in Patients Undergoing Ureterorenoscopy
Brief Title: Effects of Virtual Reality and Stress Ball on Fear, Pain, Anxiety, and Satisfaction in Ureterorenoscopy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Principal Investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TU-BOZKUL-013
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ureteroscopy
Keywords: Virtual reality; Stress ball; Anxiety; Pain; Patient satisfaction; Nursing
MeSH Terms: conditions — Anxiety Disorders; Pain; Patient Satisfaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The allocation of patients included in the study to groups will be performed by a researcher not involved in the data collection (YG) using a simple randomization method with a random number table. The table will be generated using the website https://www.randomizer.org/. When a patient scheduled for ureterorenoscopy arrives at the urology clinic, the principal investigator (GB) and researcher (ESS) will assess the patient according to the inclusion criteria. If the patient meets the inclusion criteria and signs the informed consent form, GB and ESS will inform YG, who will assign the patient to a group and notify GB of the assignment. In this way, all researchers other than YG, the patients, their relatives, and clinical staff will be blinded to group allocation. To prevent bias in statistical analyses, the data of patients whose data collection is complete will be entered into the database by YG coded as K1, K2, and K3 without specifying group names, and the analyses will be conduc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality group (Experimental): Patients in the virtual reality (VR) study group will watch videos in the clinic using a virtual reality headset. Patients will be asked to lie in a supine position and wear a VR headset (Shinecon SC-G04E Virtual Reality Headset) compatible with Android smartphones, equipped with headphones that minimize sound loss. Through the VR headset, patients will be shown nature scenes with a relaxing music background, which can be adjusted to the patient's preferred volume. After each use, the VR headset will be disinfected according to the usage instructions.
  Interventions: Other: Virtual Reality
- Stress Ball Group (Experimental): The stress ball group, patients were instructed on how to use the stress ball. After receiving the stress ball, they were asked to squeeze it up to five times every three counts. Patients were advised to continue using the stress ball until they left the clinic. Each stress ball was assigned to a single patient and not shared.
  Interventions: Other: Stress Ball
- Control group (No Intervention): In the control group, the routine pre-procedure procedures and standard clinical practices will be applied

INTERVENTIONS:
Other: Virtual Reality — Patients in the virtual reality (VR) study group will watch videos in the clinic using a virtual reality headset. Patients will be asked to lie in a supine position and wear a VR headset (Shinecon SC-G04E Virtual Reality Headset) compatible with Android smartphones, equipped with headphones that minimize sound loss. Through the VR headset, patients will be shown nature scenes with a relaxing music background, which can be adjusted to the patient's preferred volume. After each use, the VR headset will be disinfected according to the usage instructions.
  Arms: Virtual reality group
Other: Stress Ball — In the stress ball group, patients were instructed on how to use the stress ball. After receiving the stress ball, they were asked to squeeze it up to five times every three counts. Patients were advised to continue using the stress ball until they left the clinic. Each stress ball was assigned to a single patient and not shared.
  Arms: Stress Ball Group

SUMMARY:
This study aimed to determine the effects of virtual reality and stress ball interventions on procedure-related fear, anxiety, and patient satisfaction in patients undergoing ureterorenoscopy. The study is a prospective, randomized controlled clinical trial. The sample size was calculated to ensure sufficient statistical power to detect an effect size of Cohen's f = 0.333, considering α = 0.05, power (1-β) = 0.80, and number of groups = 3, resulting in 30 participants per group, for a total of 90 patients undergoing ureterorenoscopy.

Data will be collected using the "Demographic Information Form," "State Anxiety Inventory," "Procedure-Related Fear Scale," "Visual Analog Scale," and "Newcastle Satisfaction with Nursing Care Scale." Upon admission to the clinic for the procedure, all patients will complete the "Demographic Information Form," "State Anxiety Inventory," and "Procedure-Related Fear Scale" prior to the surgical intervention.

Patients in the virtual reality group will view nature scenes with relaxing music via a virtual reality headset in the clinic, with the sound level adjusted according to the patient's preference. Patients in the stress ball group will be instructed to squeeze the ball up to five counts every three counts. The control group will receive the routine pre-procedure procedures and standard care in the clinic.

After the procedure, when patients return to the clinic (and are in bed), the "State Anxiety Inventory," "Visual Analog Scale," and "Newcastle Satisfaction with Nursing Care Scale" will be administered. Data analysis will include descriptive statistics and appropriate parametric or non-parametric tests (t-test, Mann-Whitney U, Kruskal-Wallis). A p-value of <0.05 will be considered statistically significant in comparisons.

DETAILED DESCRIPTION:
This study aimed to determine the effects of virtual reality and stress ball interventions on procedure-related fear, anxiety, and patient satisfaction in patients undergoing ureterorenoscopy. The study is a prospective, randomized controlled clinical trial. The sample size was calculated to ensure sufficient statistical power to detect an effect size of Cohen's f = 0.333, considering α = 0.05, power (1-β) = 0.80, and number of groups = 3, resulting in 30 participants per group, for a total of 90 patients undergoing ureterorenoscopy. Data will be collected using the "Demographic Information Form," "State Anxiety Inventory," "Procedure-Related Fear Scale," "Visual Analog Scale," and "Newcastle Satisfaction with Nursing Care Scale." Upon admission to the clinic for the procedure, all patients will complete the "Demographic Information Form," "State Anxiety Inventory," and "Procedure-Related Fear Scale" prior to the surgical intervention.

Patients in the virtual reality group will view nature scenes with relaxing music via a virtual reality headset in the clinic, with the sound level adjusted according to the patient's preference. Patients in the stress ball group will be instructed to squeeze the ball up to five counts every three counts. The control group will receive the routine pre-procedure procedures and standard care in the clinic.

After the procedure, when patients return to the clinic (and are in bed), the "State Anxiety Inventory," "Visual Analog Scale," and "Newcastle Satisfaction with Nursing Care Scale" will be administered. The data will be analyzed using computer software. Patients' descriptive characteristics will be summarized as mean ± standard deviation, median (minimum-maximum), percentage, and frequency values. Qualitative data from the patient follow-up form will be categorized, converted into quantitative data, and presented as percentages and frequency distributions. After examining the normality of the data distribution, one-way analysis of variance (One-Way ANOVA) will be used to compare continuous variables showing a normal distribution among the three independent groups. For continuous variables that do not show a normal distribution, group comparisons will be performed using the Kruskal-Wallis H test. When a significant difference is found between groups, appropriate post-hoc analyses will be applied. The level of statistical significance will be set at p < 0.05 with a 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* • Aged 18 years or older,

  * Scheduled for ureteroscopy (URS),
  * Fully conscious, oriented, and cooperative,
  * Provided written informed consent to participate in the study,
  * Able to speak and understand Turkish,
  * Without visual or hearing impairments,
  * No prior experience with virtual reality (VR),
  * Without any mental health disorders.

Exclusion Criteria:

* Those who do not wish to participate or who wish to withdraw from the study, • Patients with chronic pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 6 months
  The State Anxiety Scale : In this study, the DAQ, which is structured to measure momentary feelings, was used. Its Turkish validity and reliability was conducted by Öner and Le Compte in 1983. The DAQ consists of 20 questions on a four-point Likert scale. The statements in the DAQ are evaluated as not at all (1), a little (2), a lot (3) and completely (4). In this section, the statements are divided into direct and reversed statements. Inverted statements: 1st, 2nd, 5th, 5th, 8th, 8th, 10th, 11th, 15th, 16th, 19th, 20th items. The total score of the reversed statements is subtracted from the total score of the direct statements and the number 50, which is the invariant value of the DAQ, is added to the value obtained and the DAQ score is calculated. The scale score ranges between 20-80 and an increase in the score indicates an increase in the level of anxiety.
Procedure-Related Pain | 6 months
  Visual Analog Scale: It is a scale that provides a subjective assessment of pain on a horizontal or vertical line from 0 (no pain at all)-10 (very severe pain) to evaluate the level of pain (Wewers and Lowe, 1990).

SECONDARY OUTCOMES:
Fear | 6 months
  Patients' fear will be assessed using a visual analog scale (VAS) ranging from 0 to 10; 0 represents "No fear at all," and 10 represents "Maximum fear." The minimum possible score is 0, and the maximum score is 10. Higher total scores indicate a higher level of fear experienced by the patient during or prior to the procedure.
Patient Satisfaction | 6 months
  Newcastle Satisfaction with Nursing Care Scale: Developed by Thomas et al. (1996), the Newcastle Satisfaction with Nursing Care Scale (NSNS) is used to assess the quality of nursing care in hospitals. The scale was adapted into Turkish by Uzun in 2003, and its validity and reliability were evaluated by Akın and Erdoğan in 2007 (Akin & Erdogan, 2007). The scale consists of 19 items rated on a five-point Likert scale, with scores ranging from 1 (Not satisfied at all) to 5 (Very satisfied). The total score reflects the level of satisfaction with nursing care (minimum: 19, maximum: 95). In the original study, the reliability coefficient was 0.96, while in the Turkish adaptation it was 0.94, and 0.96 in the subsequent validity and reliability study.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sibal NS, Sibal I, Aksoy HZ, Aydin HR, Ozoran Y, Sekerci CA. The Effect of Virtual Reality Headset Use on Anxiety Levels During Urodynamic Testing: A Prospective, Randomized Controlled Study. Urology. 2025 Dec;206:48-55. doi: 10.1016/j.urology.2025.08.002. Epub 2025 Aug 6. PMID 40780518
- [Result] Genc H, Korkmaz M, Akkurt A. The Effect of Virtual Reality Glasses and Stress Balls on Pain and Vital Findings During Transrectal Prostate Biopsy: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):344-350. doi: 10.1016/j.jopan.2021.09.006. Epub 2022 Apr 7. PMID 35397973